CLINICAL TRIAL: NCT03784846
Title: Mindfulness-Based Resilience Training for Aggression, Health, and Stress Among Law Enforcement Officers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michael Christopher, PhD, Multiple Principal Investigator, Pacific University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1295787-14; U01AT009841 (NIH)
Record Dates: First submitted 2018-12-13; First posted 2018-12-24 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Stress, Psychological; Aggression
MeSH Terms: conditions — Stress, Psychological; Aggression

STUDY DESIGN:
Intervention Model Description: Individually-Randomized Group Treatment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-Based Resilience Training (Experimental): MBRT is an 8-week program combining training in standardized mindfulness practices targeting factors that facilitate resilience, cognitive behavioral therapy (CBT), and psychoeducation. It contains experiential and didactic exercises including body scan, sitting and walking meditation, mindful movement and discussions.
  Interventions: Behavioral: Mindfulness-Based Resilience Training
- Stress Management Education (Active Comparator): SME was designed as an active control condition for other mindfulness-based intervention trials. SME uses a group-based didactic approach with modules on physiological and dietary effects of stress, time management, sleep physiology and insomnia, nutrition, exercise, stress hardiness, and factors mitigating impacts of stress.
  Interventions: Behavioral: Stress Management Education
- No Intervention Control (No Intervention): No contact control condition (other than baseline, post, and follow-up assessments)

INTERVENTIONS:
Behavioral: Mindfulness-Based Resilience Training — MBRT is an 8-week program combining training in standardized mindfulness practices targeting factors that facilitate resilience, CBT, and psychoeducation. It contains experiential and didactic exercises including body scan, sitting and walking meditation, mindful movement and discussions.
  Arms: Mindfulness-Based Resilience Training
Behavioral: Stress Management Education — SME was designed as an active control condition for other Mindfulness-Based Intervention trials. SME uses a group-based didactic approach with modules on physiological and dietary effects of stress, time management, sleep physiology and insomnia, nutrition, exercise, stress hardiness, and factors mitigating impacts of stress.
  Arms: Stress Management Education

SUMMARY:
Law enforcement officers (LEOs) are exposed to significant stressors, elevating their risk for aggression and excessive use of force, as well as mental health consequences, including post-traumatic stress disorder, burnout, alcohol misuse, depression, and suicide. The proposed study will identify, optimize and refine best clinical and research practices across two sites to ensure success in a future multisite efficacy trial assessing preventative effects of Mindfulness-Based Resilience Training on physiological, behavioral, and psychological outcomes.

DETAILED DESCRIPTION:
Law enforcement officers (LEOs) are exposed to significant stressors, elevating their risk for aggression and excessive use of force. Such dysfunctional stress reactivity can lead to devastating consequences for their community, including unjustified shootings, severe beatings, and fatal chokings. It can also lead to serious consequences for the LEOs, including elevated incidence of post-traumatic stress disorder, burnout, alcohol misuse, depression, and suicide. A recent meta-analysis of LEO stress reduction programs found little evidence to demonstrate that such approaches are effective, highlighting the urgent need for preventive interventions targeting the stress inherent to policing. Mindfulness training is a promising approach with high-stress populations that has been shown effective in reducing stress and increasing resilience. In a recent pilot feasibility study (R21AT008854), the study team established initial feasibility, acceptability, and adherence to procedures in a single-site RCT assessing Mindfulness-Based Resilience Training (MBRT), a preventive intervention designed to improve LEO mental health and resilience, and reduce aggression and excessive use of force. The R21 data suggest physiological mechanisms and potential clinical benefit in a sample of LEOs. Relative to waitlist control, MBRT participants showed improvements in stress reactivity, aggression, burnout, occupational stress, sleep disturbance, and psychological flexibility. Implemented at two sites, the proposed study is designed to establish optimal protocols and procedures for a future full-scale, multi-site trial assessing effects of MBRT versus an attention control (Stress Management Education) and a no-intervention control, on physiological, behavioral, and psychological outcomes. To prepare for this future clinical trial, this study will: a) enhance efficiency of recruitment, engagement and retention; b) optimize lab, assessment, and data management procedures; c) optimize intervention training and ensure fidelity to intervention protocols; and d) assess participant experience and optimize outcome measures across sites. The long-term objective of this line of research is to develop an intervention that will reduce violence and increase resilience among LEOs, as well as yield significant benefits for communities and residents they serve.

ELIGIBILITY:
Inclusion Criteria:

* be 21-65 years old (age limitations for both police departments),
* demonstrate English fluency,
* be a sworn, full-time, active status law enforcement officer,
* agree to random assignment to condition, and
* be willing to complete assessments at multiple time points and attend intervention groups

Exclusion Criteria:

* previous participation in MBSR, MBRT or a similar mindfulness course,
* score in the severe range on brief screening measures of depression, suicidal ideation, alcohol use, or PTSD, or
* unable or unwilling to give written informed consent.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of New Mexico, Albuquerque, New Mexico
  - Pacific University, Forest Grove, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Christopher M, Bowen S, Witkiewitz K. Mindfulness-based resilience training for aggression, stress and health in law enforcement officers: study protocol for a multisite, randomized, single-blind clinical feasibility trial. Trials. 2020 Feb 28;21(1):236. doi: 10.1186/s13063-020-4165-y. PMID 32111233
- [Derived] Christopher M, Bowen S, Witkiewitz K, Grupe D, Goerling R, Hunsinger M, Oken B, Korecki T, Rosenbaum N. A multisite feasibility randomized clinical trial of mindfulness-based resilience training for aggression, stress, and health in law enforcement officers. BMC Complement Med Ther. 2024 Apr 4;24(1):142. doi: 10.1186/s12906-024-04452-y. PMID 38575888
- [Derived] Christopher M, Ferry M, Simmons A, Vasquez A, Reynolds B, Grupe D. Psychometric properties of the Buss-Perry Aggression Questionnaire-short form among law enforcement officers. Aggress Behav. 2024 Mar;50(2):e22145. doi: 10.1002/ab.22145. PMID 38477412

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants were assigned to a study arm.
Groups:
- Mindfulness-Based Resilience Training (MBRT): MBRT is an 8-week program combining training in standardized mindfulness practices targeting factors that facilitate resilience, cognitive behavioral therapy (CBT), and psychoeducation. It contains experiential and didactic exercises including body scan, sitting and walking meditation, mindful movement and discussions.
- Stress Management Education (SME): SME was designed as an active control condition for other mindfulness-based intervention trials. SME uses a group-based didactic approach with modules on physiological and dietary effects of stress, time management, sleep physiology and insomnia, nutrition, exercise, stress hardiness, and factors mitigating impacts of stress.
Period: Pre-COVID Study
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Started | 17 | 14 | 5
Completed | 6 | 3 | 0
Not Completed | 11 | 11 | 5
Not completed — Lost to Follow-up | 3 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Discontinued by Researchers | 7 | 6 | 2
Period: Post-COVID Study
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Started | 33 | 24 | 16
Completed | 29 | 17 | 15
Not Completed | 4 | 7 | 1
Not completed — Lost to Follow-up | 3 | 5 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Resilience Training | Stress Management Education | No Intervention Control | Total
Number analyzed (Participants) | 50 | 38 | 21 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 38 | 21 | 109
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.22 (10.03) | 39.18 (8.06) | 38.90 (10.09) | 39.61 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 5 | 26
  Male | 38 | 29 | 16 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 9 | 4 | 29
  Not Hispanic or Latino | 32 | 29 | 16 | 77
  Unknown or Not Reported | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 41 | 36 | 19 | 96
  More than one race | 4 | 1 | 1 | 6
  Unknown or Not Reported | 3 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 50 | 38 | 21 | 109

OUTCOME MEASURES:

1. Primary Outcome: Change in Aggression
Description: Buss-Perry Aggression Questionnaire-Short Form. Scores range from 1-5, with higher scores indicating greater aggression.
Time Frame: baseline, post-intervention (week 8), 3-month followup, 6-month followup
Population: Numbers at post-intervention, 3-month followup, and 6-month followup reflect attrition or participants or lost to followup.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  Baseline | 1.94 (.64) | 1.67 (.45) | 1.85 (.79)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 1.72 (.48) | 1.68 (.57) | 1.98 (.82)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 1.63 (.50) | 1.58 (.37) | 1.84 (.76)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 1.57 (.46) | 1.69 (.60) | 1.78 (.66)

2. Secondary Outcome: Change in C-reactive Protein
Description: Blood spot analysis of high-sensitivity C-reactive protein.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup
Population: Numbers at post-intervention and 3-month followup reflect attrition or participants or lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale "mg/L"
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
units on a scale "mg/L"
  baseline | 1.22 (1.42) | .61 (.62) | 2.11 (2.59)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | .99 (1.26) | .80 (1.13) | 1.11 (.76)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | .90 (1.06) | .61 (2.41) | 1.66 (.58)

3. Secondary Outcome: Change in Interleukin-6
Description: Blood spot analysis of interleukin-6.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup
Population: Numbers at post-intervention and 3-month followup reflect attrition or participants or lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale "pg/mL"
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
units on a scale "pg/mL"
  baseline | .55 (.87) | .37 (.30) | .28 (.12)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | .58 (.91) | .51 (.45) | .23 (.38)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | .37 (.28) | .39 (.29) | .23 (.11)

4. Secondary Outcome: Change in Interleukin-10
Description: Blood spot analysis of interleukin-10.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup
Population: Numbers at post-intervention and 3-month followup reflect attrition or participants or lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale "pg/mL"
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
units on a scale "pg/mL"
  baseline | .27 (.27) | .28 (.20) | .16 (.08)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | .20 (.16) | .17 (.10) | .13 (.12)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | .21 (.13) | .18 (.11) | .11 (.07)

5. Secondary Outcome: Change in Tumor Necrosis Factor-alpha
Description: Blood spot analysis of tumor necrosis factor-alpha.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup
Population: Numbers at post-intervention and 3-month followup reflect attrition or participants or lost to followup.
Measure: Mean (Standard Deviation); unit: units on a scale "pg/mL"
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
units on a scale "pg/mL"
  baseline | 2.25 (.81) | 2.20 (.66) | 1.87 (.45)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 2.02 (.68) | 1.71 (.39) | 1.70 (.62)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 1.76 (.61) | 1.71 (.35) | 1.66 (.27)

6. Secondary Outcome: Change in Psychological Resilience
Description: Brief Resilience Scale. Scores range from 1-5, with higher scores indicating greater resilience.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  Baseline | 3.71 (.74) | 4.00 (.47) | 3.99 (.40)
  post-intervention: number analyzed (Participants) | 31 | 18 | 15
  post-intervention | 4.08 (.65) | 4.11 (.49) | 3.90 (.67)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 3.98 (.72) | 4.10 (.41) | 4.03 (.41)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 4.04 (.66) | 4.01 (.52) | 3.83 (.67)

7. Secondary Outcome: Change in Alcohol Use
Description: Patient Reported Outcome Measurement System (PROMIS) Alcohol Use. Scores range from 39-77, with higher scores indicating greater alcohol use.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 46.62 (7.48) | 45.50 (7.46) | 44.42 (5.79)
  post-intervention (8 weeks): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (8 weeks) | 46.95 (7.60) | 48.54 (6.58) | 45.73 (6.50)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 48.00 (7.72) | 49.01 (6.51) | 45.78 (6.20)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 47.82 (6.82) | 46.65 (7.74) | 48.98 (5.94)

8. Secondary Outcome: Change in Alcohol Use Negative Consequences
Description: Patient Reported Outcome Measurement System (PROMIS) Alcohol Use Negative Consequences.Scores range from 39-77, with higher scores indicating greater alcohol use negative consequences.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 40.67 (5.44) | 40.35 (5.21) | 40.49 (4.91)
  post-intervention (8 weeks): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (8 weeks) | 40.98 (4.99) | 41.06 (5.35) | 41.03 (4.80)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 40.81 (5.40) | 41.06 (4.93) | 42.53 (5.47)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 41.26 (5.17) | 40.81 (5.34) | 40.74 (5.51)

9. Secondary Outcome: Change in Depression
Description: Patient Reported Outcome Measurement System (PROMIS) Depression. Scores range from 38-80, with higher scores indicating more depression.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 50.15 (7.99) | 48.17 (6.69) | 48.22 (7.56)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 49.22 (5.74) | 48.02 (8.66) | 47.55 (9.17)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 49.50 (7.36) | 49.01 (7.87) | 47.13 (5.93)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 48.98 (7.35) | 48.14 (8.07) | 46.73 (9.49)

10. Secondary Outcome: Change in Suicidal Thinking
Description: Concise Heath Risk Tracking Scale-Self-Report. Scores range from 7-35, with higher scores indicating greater suicidal ideation.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 8.91 (2.39) | 8.16 (2.23) | 8.20 (2.65)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 8.74 (2.67) | 8.05 (2.25) | 9.57 (4.18)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 8.90 (3.34) | 8.58 (2.62) | 8.27 (1.98)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 8.07 (1.73) | 8.44 (2.64) | 8.21 (2.19)

11. Secondary Outcome: Change in Trauma Symptoms
Description: PTSD Checklist for DSM-5. Scores ranges from 0-80, with higher scores indicating greater PTSD symptoms.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 37.76 (14.39) | 33.36 (9.12) | 31.53 (12.13)
  post-intervention (week 8) | 34.32 (11.69) | 30.74 (8.77) | 33.36 (15.35)
  3-month followup | 34.07 (12.57) | 32.29 (10.26) | 33.20 (11.94)
  6-month followup | 31.93 (11.74) | 31.61 (11.08) | 32.07 (13.09)

12. Secondary Outcome: Change in Burnout
Description: Oldenburg Burnout Inventory. Scores range from 1-4, with higher scores indicating greater burnout.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 2.40 (.46) | 2.36 (.35) | 2.38 (.36)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 2.39 (.44) | 2.36 (.29) | 2.33 (.26)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 2.34 (.38) | 2.33 (.30) | 2.36 (.24)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 2.32 (.42) | 2.42 (.35) | 2.37 (.28)

13. Secondary Outcome: Change in Sustained Attention
Description: Sustained Attention to Response Task. A computer-based go/no-go task that requires participants to withhold behavioral response to a single, infrequent target presented amongst a background of frequent non-targets. Increased errors indicates less sustained attention.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
errors
  baseline | 17.03 (13.50) | 16.00 (53.10) | 31.42 (37.16)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 15.86 (30.28) | 13.50 (20.00) | 30.71 (30.01)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 15.33 (18.88) | 9.30 (11.06) | 25.35 (20.48)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 15.88 (27.22) | 9.53 (6.89) | 29.23 (63.90)

14. Secondary Outcome: Change in Perceived Stress
Description: Perceived Stress Scale-10. Scores range from 0-40, with higher scores indicating greater perceived stress.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 24.45 (6.13) | 23.16 (4.60) | 22.93 (6.52)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 23.39 (5.71) | 22.05 (4.39) | 22.86 (7.37)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 22.66 (6.61) | 23.65 (5.90) | 22.47 (7.26)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 22.97 (6.31) | 24.00 (4.23) | 23.00 (5.48)

15. Secondary Outcome: Change in Sleep Disturbance
Description: Patient Reported Outcome Measurement System (PROMIS) Sleep Disturbance. Scores range from 32-76, with higher scores indicating greater sleep disturbance.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 54.35 (7.32) | 52.48 (7.80) | 53.48 (9.88)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 52.03 (7.72) | 54.38 (6.44) | 53.11 (9.26)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 51.45 (7.87) | 52.93 (7.65) | 53.85 (7.97)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 51.36 (6.62) | 51.51 (7.78) | 52.90 (9.79)

16. Secondary Outcome: Change in Self-Compassion
Description: Self-Compassion Scale-Short Form. Scores range from 1-5, with higher scores indicating greater self-compassion.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 3.35 (.66) | 3.52 (.58) | 3.16 (.73)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 3.52 (.64) | 3.54 (.59) | 3.40 (.83)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 3.61 (.57) | 3.56 (.52) | 3.41 (.76)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 3.66 (.53) | 3.45 (.55) | 3.38 (.76)

17. Secondary Outcome: Change in Mindfulness
Description: Five Facet Mindfulness Questionnaire-Short Form. Scores range from 1-5, with higher scores indicating greater mindfulness.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 3.48 (.68) | 3.53 (.47) | 3.63 (.74)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 3.56 (.45) | 3.61 (.41) | 3.56 (.84)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 3.60 (.60) | 3.51 (.29) | 3.65 (.58)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 3.62 (.45) | 3.51 (.45) | 3.61 (.64)

18. Secondary Outcome: Change in Interoceptive Awareness
Description: Multidimensional Assessment of Interoceptive Awareness-II. Scores range from 1-6, with higher scores indicating greater interoceptive awareness.
Time Frame: baseline, post-intervention (8 weeks), 3 month followup, 6 month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale
  baseline | 3.89 (.64) | 3.77 (.61) | 3.62 (.51)
  post-intervention (week 8): number analyzed (Participants) | 31 | 18 | 15
  post-intervention (week 8) | 4.19 (.50) | 3.82 (.52) | 3.89 (.55)
  3-month followup: number analyzed (Participants) | 29 | 16 | 16
  3-month followup | 4.22 (.61) | 4.00 (.50) | 3.67 (.66)
  6-month followup: number analyzed (Participants) | 29 | 17 | 15
  6-month followup | 4.19 (.55) | 3.87 (.79) | 3.62 (.59)

19. Secondary Outcome: Treatment Acceptability
Description: Postcourse satisfaction survey. Scores range from 4-16, with higher scores indicating greater treatment acceptability. Measure only administered to Mindfulness-Based Resilience Training and Stress Management Education arms.
Time Frame: post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME)
Number analyzed (Participants) | 31 | 18
score on a scale | 13.94 (2.43) | 12.28 (2.52)

20. Secondary Outcome: Treatment Compliance
Description: Objective assessment of duration of homework practice. Measure only administered to Mindfulness-Based Resilience Training and Stress Management Education arms.
Time Frame: post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME)
Number analyzed (Participants) | 31 | 18
minutes | 211.66 (186.62) | 65.45 (68.45)

21. Secondary Outcome: Treatment Expectancy and Credibility
Description: Expectancy/Credibility Questionnaire. Scale for measuring treatment expectancy and rationale credibility for use in clinical outcome studies. Scores range from 7-21, with higher scores indicating greater expectancy and credibility.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME) | No Intervention Control
Number analyzed (Participants) | 33 | 24 | 16
score on a scale | 15.61 (3.75) | 15.60 (2.90) | 15.53 (2.20)

22. Secondary Outcome: Global Impression of Change
Description: Clinical Global Impressions Scale. Measure of perceived change in functioning as a result of the intervention. Scores range from 3-21, with higher scores indicating a greater impression of change. Measure only administered to Mindfulness-Based Resilience Training and Stress Management Education arms.
Time Frame: post-intervention (8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness-Based Resilience Training (MBRT) | Stress Management Education (SME)
Number analyzed (Participants) | 31 | 18
score on a scale | 16.19 (2.10) | 14.22 (1.66)

ADVERSE EVENTS:
Time Frame: The adverse event was followed for 6 months.
Arm/Group | Mindfulness-Based Resilience Training | Stress Management Education | No Intervention Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/38 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/38 | 0/21
Other Adverse Events (participants affected / at risk) | 1/50 | 0/38 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness-Based Resilience Training (N=50) | Stress Management Education (N=38) | No Intervention Control (N=21)
Participant contracted COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: pre-COVID (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT03784846/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: post-COVID (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT03784846/Prot_SAP_002.pdf
  • Informed Consent Form (2021-03-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT03784846/ICF_000.pdf